CLINICAL TRIAL: NCT06015542
Title: Self-administration of Subcutaneous Elranatamab in the Patients' Homes. An Open Label, Phase Two, Prospective, Multi-center, Non-randomized, Sponsor-initiated Explorative Trial
Brief Title: Self-administration of Subcutaneous Elranatamab in the Patients' Homes.
Acronym: ERICA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Lund (Other)
Collaborators: Pfizer (Industry); Vejle Hospital (Other)
Responsible Party: Sponsor-Investigator, Thomas Lund, Principal Investigator, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERICA
Record Dates: First submitted 2023-08-21; First posted 2023-08-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: An open label, phase two, prospective, multi-center, non-randomized, sponsor-initiated explorative trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Self-administration of Elranatamab (Experimental): It is a feasibility study assessing the feasibility and safety of self-administration of Elranatamab in the homes of the patients. The intervention of the study is self-administration of Elranatamab by the patient, thereby changing the administration from an outpatient setting to a home setting. The patients will function as their own controls, as treatment will be given alternately at home and in the outpatient clinic.
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — Elranatamab will be administered as monotherapy for six cycles of 28 days. Elranatamab 76 mg will be administered QW with a 2-step-up priming dose regimen administered during the first week (12 mg D1 and 32 mg D4).
  Other Names: PF-06863135

SUMMARY:
The goal of this open label, phase two, prospective, non-randomized, sponsor-initiated explorative trial is to test self-administration of subcutaneous Elranatamab in the patients' homes in patients with relapsed multiple myeloma exposed to at least one proteasome inhibitor, one IMID and one anti CD-38 antibody. The main question[s]it aims to answer are:

* To evaluate the safety of self-administration of Elranatamab in the patients' own homes using registrations of occurrence of CRS, Immune effector cell-associated neurotoxicity syndrome (ICANS) and infections.
* To evaluate the feasibility of self-administration of Elranatamab in the patients´ own homes by registration of discarded doses, planned doses administered at home and doses diverted from the patients' homes to the outpatient clinic.
* To elucidate the perspectives of patients and their caregivers of self-administration of Elranatamab at home by interviewing both parties at end of treatment (EOT).
* To elucidate the perspectives of involved healthcare professionals in a focus group interview at end of study (EOS).
* To clarify time spent on self-administration at home compared to administration at the outpatient clinic by registering time consumption for patients, caregivers and healthcare professionals.
* To evaluate the patients' QoL during self-administration using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) together with the Functional Assessment of Cancer Therapy-Cognitive (FACT Cognitive).
* To clarify if self-administration in the patients' homes leads to additional unplanned contacts with the healthcare system as a whole by weekly registration of any unplanned contacts.
* To determine financial costs of self-administration at home compared to administration at the outpatient clinic from the perspectives of patients, caregivers and the healthcare system by collecting data on lost earnings, transport costs and salary costs.
* To evaluate the feasibility of the use of an electronic registration of side effects prior to treatment by comparing electronic patient reported outcome (PRO) data to registrations performed by nurses in the outpatient clinic during telephone consultations.

Participants will be asked to

* register time spend
* answer PRO-questionnaires
* weekly register any unplanned contact to the heathcare system
* be interviewed

DETAILED DESCRIPTION:
Background Bispecific antibodies targeting CD3 and BCMA have demonstrated astonishing efficacy with response rates of nearly 65 % in triple class exposed patients with multiple myeloma (MM). This will not necessarily be the first product to be marketed, but might be a product proven to be applicable for safe and convenient self-administration in the patients' homes, thereby improving the patients' and their caregivers' Quality of Life (QoL) and reducing the burden on the healthcare system. Although optimal dosing regimens are still being investigated, most CD3xBCMA are given weekly until progression, with the possibility of downscaling to twice monthly, if good remission is obtained. Consequently, patients have multiple visits to the outpatient clinic, meaning that they spend a substantial amount of time on transport, and that they are continuously exposed to potential infections. Furthermore, the outpatient clinic might end out with many bispecific treatments in the future, due to their high efficiency, thus straining the logistics of the hospital.

Previous studies have shown that patients who administer their treatment themselves experience better QoL, a higher level of well-being, and have a higher level of daily activity. In addition, socio-economic savings of up to 20-50% are seen with self-administration compared to outpatient treatment.

Elranatamab is a bispecific CD3xBCMA with some unique properties; it is given subcutaneously as a fixed dose, and it has shown a remarkably low risk of CRS after the third injection. This makes it a perfect candidate to investigate in a setup, where patients are trained in self-administration at their own homes.

Acquiring source data and planned visits In the study, Elranatamab will be administered as monotherapy for six cycles of 28 days (Table 1). Patients will receive subcutaneous Elranatamab 76 mg QW with a 2-step-up priming dose regimen administered during the first week (12 mg D1 and 32 mg D4). For safety reasons, the step-up doses will be administered with hospitalization for a minimum of 48hr (C1D1) and 24hr (C1D4), respectively. During hospitalization, vital signs will be measured at least 6 times per overnight stay. If treatment is tolerated, C1D8, C1D15 and C1D22 will be administered in the outpatient clinic and will include training of the patients in self-administration. In cycle 2 to cycle 6, patients will administer the treatment themselves in the outpatient clinic D1 and at home D8, D15 and D22. However, if patients experience any CRS during the study, the consecutive two doses must be administered in the outpatient clinic without any signs of CRS, before home treatment can be resumed. If patients experience ICANS, they will be taken off study.

Prior to each new treatment cycle, laboratory assessments will be conducted at the local hospital or at the patient's GP, according to general standards. A hematologist at Odense University Hospital, who will also evaluate the patient, must accept the laboratory assessments before D1 of all cycles.

Further, the following data will be collected to meet the secondary endpoints:

At inclusion, data on age, gender, marital status, PS, R-ISS, ISS, vital signs, myeloma type, renal and liver function, concomitant medication (CM), weight, number of previous lines of treatment and response to previous lines of treatment will be registered in an electronic case report form (eCRF). Further, patients will be physically examined and cognitively tested, which will include a writing test and a test of their ability to recognize known pictures. Finally, patients must complete the EORTC QLQ-C30 and the FACT Cognitive questionnaires electronically.

During planned hospitalization in cycle 1, patients will be continuously examined, and data on PS, vital signs, results of blood samples, CM, AEs and results of CRS and ICANS screening will be collected. Similar data will be collected at C1D8, C1D15 and C1D22.

Starting from cycle 2, data on location of administration will be collected. Specifically, redirected administrations and discarded doses will be registered. When patients show in the outpatient clinic at D1, they will be physically examined, and data on PS, vital signs, results of blood samples, CM, AEs, weight and result of CRS and ICANS screening will be collected. Further, patients should complete the EORTC QLQ-C30 electronically. If they do not complete the questionnaire during their visit at the outpatient clinic, it can be completed from home the following days, but no later than two days after treatment (D3).

Before each home administration (D8, D15 and D22), patients will receive an electronic questionnaire on their physical and cognitive condition. They must answer if they have had a fever (they will be instructed in measuring their temperature before every injection), dizziness or any other sickness, or if they have received any antibiotics since their last administration. Further, to rule out any grade of ICANS, they will be cognitively tested. The questionnaire must be filled in within two days prior to the administration. On the day of treatment, a specialized nurse from the outpatient clinic will assess the responses and call the patient in the morning to make sure there are no unexpected problems or fever, which would be incompatible with treatment.

At D1 (in the outpatient clinic) and D8 (at home) in cycle 2-6, patients, caregivers, nurses and physicians in the outpatient clinic must register their time spent on the administration. For patients and caregivers, this includes waiting time and time spent on transportation. Further, they should register their mode of transportation and if they have had any need for taking time off from work due to the planned administration. For nurses and physicians, this includes both administrative and time spent with the patient.

Throughout the study, patients must register if they have had any unplanned contact with the healthcare system (e.g. to with the Department of Hematology or their GP). For this purpose, they will automatically be contacted electronically each week, and if they register any unplanned contacts, a study nurse will contact them for clarification and register the cause of the contact.

At EOT, patients and caregivers must complete a questionnaire on their preferences (treatment at home or in the outpatient clinic). Moreover, patients must complete the EORTC QLQ-C30 and FACT Cognitive questionnaires. Finally, patients and caregivers will be interviewed individually.

At EOS, a focus group interview with involved health care professionals at the outpatient clinic will be conducted.

Safety considerations and drug administration The most common AE associated with Elranatamab is CRS. The treatments in the first cycle will be administered at the hospital; the two priming doses with hospitalization and the others in the outpatient clinic. Further, to reduce the grade of CRS, patients will receive premedications including corticosteroid, antihistamine and antipyretic for both priming doses and for the first full dose. If no CRS is observed, only antihistamine and antipyretic will be used in the following treatments. Treatment will not be released for self-administration before cycle 2, at which time the risk of severe CRS is considered minimal. Further, to reduce the risk of infections, patients will receive infection prophylaxis in the form of Sulfametoxazole with Trimethoprim 80/400mg daily, Ciprofloxacin 500mg twice daily, as well as immunoglobulin substitution, if polyclonal IgG drops below 5 g/L.

Before each new treatment cycle is initiated, laboratory assessments will be conducted at the local hospital or the patient's GP, according to general standards. A hematologist at Odense University Hospital, who will also evaluate the patient, must accept the laboratory assessments before treatment is released. Before each home administration (D8, D15 and D22), the patient must answer an electronic questionnaire on their physical and cognitive condition. This includes questions on whether they have had a fever, dizziness or any other sickness, and if they have received any antibiotics since last their last administration). Further, to rule out any grade of CRS or infection, patients will be instructed in measuring their temperature before every injection and report the result electronically. Finally, to rule out any grade of ICANS, they will be cognitively tested, which will include a writing test and a test of their ability to recognize known pictures.

At the day of administration, a specialized nurse will assess the responses and call the patient in the morning to make sure no unexpected problems or fever have occurred. If all criteria are met, the nurse will contact the Hospital Pharmacy that will prepare the treatment and send it directly to the patient by car.

CRS and ICANS Management of CRS and ICANS will be handled as per local guideline following ASTCT guidelines.

If the patients experience CRS (any grade) at any time, the patients must receive the two consecutive doses under observation at the hospital. Patients experiencing ICANS (any grade) will be excluded from the study.

Side effects Registration and reporting of AE, SAE and SUSAR All protocol registered AEs, SAEs and product quality complaints, whether serious or non-serious, related or not related, collected as per national guidelines to the licensed medical holder (©Pfizer) will be registered in the eCRF. SAEs will be assessed by PI as either Suspected Adverse Reaction (SAR), Suspected Unexpected Serious Adverse Reactions (SUSAR) or non-related SAE. SARs and SUSARs will be reported to the medical license holder within 24 hours of investigator acknowledgement using the Investigator Sponsored Research or Clinical Research Collaboration Interventional Study Serious Adverse Event Form V. 5.0. The form can be completed by a study coordinator, but should be signed by PI (MD. PhD, Thomas Lund) as soon as possible. However, the signature should not delay submission of the form beyond the 24 hours.

Non-related SAEs and AEs will be reported every third month to Pfizer and annually to the Danish Medical Agency.

Side effects Registration and reporting of AE, SAE and SUSAR All protocol registered AEs, SAEs and product quality complaints, whether serious or non-serious, related or not related, collected as per national guidelines to the licensed medical holder (©Pfizer) will be registered in the eCRF. SAEs will be assessed by PI as either Suspected Adverse Reaction (SAR), Suspected Unexpected Serious Adverse Reactions (SUSAR) or non-related SAE. SARs and SUSARs will be reported to the medical license holder within 24 hours of investigator acknowledgement using the Investigator Sponsored Research or Clinical Research Collaboration Interventional Study Serious Adverse Event Form V. 5.0. The form can be completed by a study coordinator, but should be signed by PI (MD. PhD, Thomas Lund) as soon as possible. However, the signature should not delay submission of the form beyond the 24 hours. The SAE form should be sent to the following password-protected e-mail: DNK.AEReporting@pfizer.com Non-related SAEs and AEs will be reported every third month to Pfizer and annually to the Danish Medical Agency.

The NCI CTCAE v 4.0 is used for grading the severity of AEs. Each dose modification or treatment delay, as well as the reason will be documented in the eCRF. AEs and SAEs will be registered from first dose of treatment until 28 calendar days after the last dose of Elranatamab in the study. In addition, any AE/SAE occurring after the 28-day period will also be registered, if PI suspects a causal relationship between Elranatamab and the AE/SAE. Signs or symptoms directly related to MM or planned hospitalization for earlier known diseases will not be registered.

ELIGIBILITY:
Inclusion criteria

* ≥ 18 years of age at the time of signing the informed consent form.
* Relapsed MM according to the IMWG criteria.
* Measurable disease defined as: M-protein quantities ≥ 0.5 g/dL by serum protein electrophoresis (sPEP) or ≥ 200 mg/24-hour urine collection by urine protein electrophoresis (uPEP) and/or Serum free light chain (FLC) levels > 100 mg/L (10 mg/dL) involved light chain and an abnormal kappa/lambda (κ/λ) ratio in patients without measurable disease in the serum or urine.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0, 1 or 2.
* Previously exposed to at least two of the following; one proteasome inhibitor, one IMID, or one anti CD-38 antibody.
* Documented disease progression during or after last anti-myeloma regimen.
* Possibility of being observed by a capable caregiver during self-administration.
* ANC ≥1.0 x 109/L (G-CSF allowed).
* Platelets ≥25 x 109/L.
* Female patients of childbearing potential must have a negative serum pregnancy test at screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.

Exclusion Criteria:

* Any significant medical condition, laboratory abnormality or psychiatric illness that would prevent the subject from participating in the study.
* Prior history of ICANS.
* Prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years with the exception of the following non-invasive malignancies:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes and metastasis] clinical staging system) or prostate cancer that is curative
* Plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes) or clinically significant Amyloidosis.
* Female who is pregnant, breastfeeding or who intends to become pregnant during the participation in the study.
* Positivity for human immunodeficiency virus (HIV), chronic or active hepatitis B or active hepatitis A or C.
* Resident on an unbridged island.
* Not being able to register PRO-data electronically.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of self-administration of Elranatamab in the patients' own homes assessed by checklist | approximately 24 weeks
  Registrations of occurrence of CRS, Immune effector cell-associated neurotoxicity syndrome (ICANS) and infections.

SECONDARY OUTCOMES:
evaluate the feasibility of self-administration of Elranatamab in the patients´ own homes | approximately 24 weeks
  registration of discarded doses, planned doses administered at home and doses diverted from the patients' homes to the outpatient clinic.
elucidate the perspectives of patients and their caregivers of self-administration of Elranatamab at home | approximately 1 hour
  interviewing both parties at end of treatment (EOT).
elucidate the perspectives of involved healthcare professionals | approximately 2 hours
  performing a focus group interview at end of study (EOS).
clarify time spent on self-administration at home compared to administration at the outpatient clinic | approximately 24 weeks
  registering time consumption for patients, caregivers and healthcare professionals.
evaluate the patients' QoL during self-administration | approximately 24 weeks
  using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) together with the Functional Assessment of Cancer Therapy-Cognitive (FACT Cognitive).
clarify if self-administration in the patients' homes leads to additional unplanned contacts with the healthcare system as a whole | approximately 24 weeks
  weekly registration of any unplanned contacts.
determine financial costs of self-administration at home compared to administration at the outpatient clinic from the perspectives of patients, caregivers and the healthcare system | approximately 24 weeks
  collecting data on lost earnings, transport costs and salary costs
evaluate the feasibility of the use of an electronic registration of side effects prior to treatment | approximately 24 weeks
  comparing electronic patient reported outcome (PRO) data to registrations performed by nurses in the outpatient clinic during telephone consultations.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lund, MD, Principal Investigator — Odense Universitetshospital
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense
  - Department of Heamatology, Vejle

IPD SHARING:
Plan to Share IPD: No
The study population is a relatively small patient group. Rewieling of IPD will potentially be a risk to human rights.